CLINICAL TRIAL: NCT00259415
Title: Evaluation of Professionally Led Support Groups for Caregivers
Brief Title: Telesupport: Evaluation of Professionally Led Support Groups for Caregivers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: IIRG-00-1998
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Caregiver Burden
Keywords: Support groups; Alzheimer's Disease
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease

INTERVENTIONS:
Behavioral: Caregiver support via telephone

SUMMARY:
This study is a collaborative effort between a community-based service organization, Supportive Older Women's Network (SOWN), and an academic research division at Thomas Jefferson University (TJU). We plan to use a randomized controlled two-group design to: 1) test the effectiveness of the intervention at 6 months to enhance social support and perceived efficacy in comparison to a control group; 2) test if gains are sustained over 12 months (within experimental group comparison); and 3) evaluate the cost and cost effectiveness of the intervention. Three secondary study aims are to describe the process and content of tele-support groups (dose/intensity, support group topics); evaluate the relative benefits for African American and White females; and determine if control group subjects benefit from receiving a peer's telephone number for mutual support (within group comparison between 6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Caregivers will be recruited for study participation who fit the following criteria: 1) female, 2) 55 or older, 3) has been a caregiver for a minimum of 6 months, 3) provides care to a person with a physician's diagnosis of ADRD, 4) has weekly access to a telephone for one hour without interruption during working hours, or if unable to have uninterrupted time, willing to have home-maker service. Homemaker service during the tele-group meetings will be arranged by the recruitment source. For this study, we plan to recruit only females since they represent the majority of those providing care to persons with ADRD and have been shown to demonstrate significantly more stress and negative health outcomes than male caregivers.

Exclusion Criteria:

* Male
* under age of 55
* not a caregiver of person with ADRD

Min Age: 55 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2000-09

PRIMARY OUTCOMES:
Caregiver depression
Caregiver burdern
Caregiver social support

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, Ph.D, Principal Investigator — Thomas Jefferson
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States